CLINICAL TRIAL: NCT05940376
Title: Efficacy and Safety of Topical Insulin in Acute-onset Neurotrophic Keratopathy After Diabetic Vitrectomy
Brief Title: Topical Insulin in Neurotrophic Keratopathy After Diabetic Vitrectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Taher Eleiwa, Professor, Benha University
Other Study IDs: RC-7-2023
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Corneal Ulcer; Neurotrophic Corneal Ulcer; Diabetes Mellitus
MeSH Terms: conditions — Corneal Ulcer; Diabetes Mellitus | interventions — Insulin, Short-Acting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Group A was assigned to receive preservative-free lubricants and prophylactic antibiotics.
- Study: Group B was assigned to receive topical insulin [1 unit per drop] 4 times per day (QID) in addition to previous treatment.
  Interventions: Drug: rapid acting insulin

INTERVENTIONS:
Drug: rapid acting insulin — Topical insulin drops were prepared by diluting 1 unit of fast-acting insulin per 1 mL of an artificial tear with a propylene glycol base. Drops were preserved at low temperature (2°C) and, was provided by the cornea specialist and was self-administered by patients at a dosage of 1 eye drop 4 times daily. Treatment continued until NK healed and then tapered accordingly. Patients would discontinue topical insulin if the condition did not improve or worsen within 4 weeks. Patients were followed up daily and slit-lamp photographs were captured with and without fluorescein corneal staining.
  Groups: Study

SUMMARY:
Various treatment options have been proposed in managing NK such as preservative-free lubrication (PF-L), withdrawal of epitheliotoxic medication, prophylactic antibiotics, applying of bandage contact lenses, using hemoderivatives 8, topical insulin, recombinant nerve growth factor (rNGF) or epidermal growth factor (rEGF).11,12, amniotic membrane transplant (AMT), or corneal neurotization.2,4,9,10 Topical insulin has been reported to effectively promote the healing of persistent corneal epithelial defects.

In our retrospective study, we explored the safety and efficacy of topical insulin, as a first-line treatment, in treatment-naïve acute NK after diabetic vitrectomy.

DETAILED DESCRIPTION:
Corneal nerves play a vital role in maintaining the homeostasis of the ocular surface. Not only mediating sensory reflexes such as blinking and lacrimation, but also corneal nerves critically maintain the integrity of corneal epithelium and the nerves themselves via producing trophic factors. An insult anywhere from the trigeminal nerve nucleus to the terminal nerve endings of the nasociliary nerve can disrupt this homeostasis and lead to corneal hypoesthesia and neurotrophic keratopathy (NK). The pathogenesis of NK has been associated with infectious, inflammatory, toxic, and iatrogenic etiologies such as ocular herpetic infection, ocular or neurologic surgery, trauma, chemical burn, diabetes, and dry eye disease. 3,4 In diabetic keratopathy, several corneal changes have been reported including abnormal basement membrane structure, poor epithelial adherence, hypothesia and alterations in the corneal stroma, Descemet membrane, and corneal endothelium. Also, NK has been reported as a rare complication of endolaser panretinal photocoagulation (PRP) and transscleral cyclophotocoagulation.7, 8, 9, 10, 11 The suggested mechanism entails the occurrence of thermal injury to the long ciliary nerve branches as they enter the suprachoroidal space at the positions corresponding to 3 and 9 o'clock on the eye. In diabetic patients, NK may present as a persistent epithelial defect refractory to conventional measures, predisposing to microbial keratitis, and/or stromal melting/scarring with subsequent perforation/blindness.3,4 Thus, rapid corneal re-epithelialization is needed to restore the corneal surface integrity.

Various treatment options have been proposed in managing NK such as preservative-free lubrication (PF-L), withdrawal of epitheliotoxic medication, prophylactic antibiotics, applying of bandage contact lenses, using hemoderivatives 8, topical insulin, recombinant nerve growth factor (rNGF) or epidermal growth factor (rEGF).11,12, amniotic membrane transplant (AMT), or corneal neurotization.2,4,9,10 Topical insulin has been reported to effectively promote the healing of persistent corneal epithelial defects.

In our study, we explored the safety and efficacy of topical insulin, as a first-line treatment, in treatment-naïve acute NK after diabetic vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult diabetic patients (18 years of age) with neurotrophic keratopathy developing within 21 days after diabetic vitrectomy. NK was classified as stage 1 (epithelial changes only without epithelial defect), stage 2 (persistent epithelial defect) or stage 3 (corneal ulcer) according to published criteria.
* decreased corneal sensitivity within the corneal lesion and in at least 1 corneal quadrant outside the lesion.

Exclusion Criteria:

* Those patients who needed intraoperative epithelial debridement during vitrectomy, having past history of ocular surgeries other than cataract surgery, or history of herpetic eye disease or limbal stem cell deficiency were excluded.
* active ocular infection or inflammation unrelated to neurotrophic keratopathy, lagophthalmos, and other ocular disease or severe vision loss in the affected eye(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult diabetic patients (18 years of age) with neurotrophic keratopathy developing within 21 days after diabetic vitrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
time to epithelial healing | 4 weeks
  healed ulcer is defined as <0.5 mm of fluorescein staining in the greatest dimension of the lesion area.

SECONDARY OUTCOMES:
any adverse effect of topical insulin or need for amniotic membrane transplantation | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study data will be available upon request
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Result] Soares RJDSM, Arede C, Sousa Neves F, da Silva Fernandes J, Cunha Ferreira C, Sequeira J. Topical Insulin-Utility and Results in Refractory Neurotrophic Keratopathy in Stages 2 and 3. Cornea. 2022 Aug 1;41(8):990-994. doi: 10.1097/ICO.0000000000002858. Epub 2021 Sep 3. PMID 34483270
- [Result] Galvis V, Nino CA, Tello A, Grice JM, Gomez MA. Topical insulin in neurotrophic keratopathy after resection of acoustic neuroma. Arch Soc Esp Oftalmol (Engl Ed). 2019 Feb;94(2):100-104. doi: 10.1016/j.oftal.2018.06.003. Epub 2018 Jul 17. English, Spanish. PMID 30025986